CLINICAL TRIAL: NCT01209611
Title: Phase 1/2 Study of Autologous Bone Marrow-Derived Mononuclear Cell Transplantation in Accelerating Soft Tissue Expansion
Brief Title: Autologous Bone Marrow-Derived Mononuclear Cell Transplantation in Accelerating Tissue Expansion and Skin Regeneration
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing-Feng Li, MD, PhD, Professor, Head of the Department of Plastic and Reconstructive Surgery, Shanghai 9th People'sHospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30730092
Record Dates: First submitted 2010-09-02; First posted 2010-09-27 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Tissue Expansion;; Skin Regeneration;; Reconstruction;; Bone Marrow Mononuclear Cells

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Autologous bone marrow mononuclear cells (Experimental): Patients received autologous MNC transplantation. Bone marrow aspirates are harvested from the anterior iliac crest of the patients under general or local anesthesia. MNCs are isolated by density gradient centrifugation. The cell suspension was adjusted to a final volume of 6-20 ml with saline. The cell suspension was injected into expanded skin intradermally via a 27-gauge needle (approximately 0.5-1×10^6 cells/cm2).
  Interventions: Procedure: Autologous bone marrow mononuclear cells
- Saline (Placebo Comparator): Patient has intradermally and subcutaneously injection of saline.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Autologous bone marrow mononuclear cells — Autologous bone marrow-derived mononuclear cells, after isolated by density gradient centrifugation from bone marrow aspiration and resuspended in saline, will be transplanted subcutaneously to expanded skin. The number of infused cells will be 1x10e6/cm2.
  Arms: Autologous bone marrow mononuclear cells
Procedure: Placebo — Patients will have mimical bone marrow aspiration under local anesthesia following with saline injection to expanded skin.
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluating whether autologous bone marrow mononuclear cells transplantation is safe and/or effective to accelerating skin regeneration and soft tissue expansion.

DETAILED DESCRIPTION:
Reconstruction of large scale skin defect is a challenge to clinical surgeons. Soft tissue expansion has won wide attention in recent years as it promotes skin regeneration with perfectly matched tissue. However, some patients with poor skin regenerative ability would suffer from skin flap over-thinned and even necrosis under the continuous stretching by silicone expander. Although, on some occasions, decelerating the expander inflation process could reduce the incidence of necrosis, this prolonged therapy circle is to be accompanied with increased complications, including infection and expander rupture, as well as the increased economic expenses by the longer hospitalization. This study is to observe the effects of autologous bone marrow mononuclear cell transplantation on accelerating skin regeneration and promoting tissue expansion process.

Patients aged between 18 to 60 years old who appear with deteriorated expanded skin will be enrolled and randomized into two groups, named as the experimental group and the control group. Patients from the experimental group will have a bone marrow aspiration and intradermal mononuclear cells transplantation. On the other side, Patients from the control group will have saline injection.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 60 years;
* Expanding skin donor site at the face, neck, anterior chest wall, abdominal wall or back;
* Implanted silicone expander of 80 to 600 ml in size;
* History of deterioration in the expanded skin texture that did not improve after the inflation procedure was suspended for more than 2 weeks;
* Persistent high level of expander internal pressure;
* Need for further skin expansion;

Exclusion Criteria:

* Not fit for soft tissue expansion treatment;
* Evidence of infection, ischemia, ulcer or other pathological changes within the targeting area which defined as not suitable for expansion; or history of delayed healing, radiational therapy;
* Significant renal, cardiovascular, hepatic and psychiatric diseases;
* Significant medical diseases or infection (including but not limited to the carrier of hepatitis B virus or HIV)
* BMI >30;
* History of any hematological disease, including leukopenia , thrombocytopenia, or thrombocytosis;
* History of allogenic bone marrow transplantation;
* Long history of smoking;
* Evidence of malignant diseases or unwillingness to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Occurence of major adverse events | Up to approximately 24 months after study start
  Including expanded flap ischaemia, necrosis, fluidify, infection, and all other adverse events
To measure inflation volume of the silicone expander | baseline, 4 weeks and 8 weeks post treatment

SECONDARY OUTCOMES:
To measure the size of expanded flap | baseline and 8 weeks post treatment
To measure the texture of expanded flap | 4 weeks and 8 weeks post treatment
To measure expanded skin thickness by ultrasound scanning | baseline, 4 weeks and 8 weeks post treatment
Laboratory examinations including routine blood test, liver function and renal function | baseline and 8 weeks post stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Qingfeng Li, MD, PhD, Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhou SB, Zhang GY, Xie Y, Zan T, Gan YK, Yao CA, Chiang CA, Wang J, Liu K, Li H, Zhou J, Yang M, Gu B, Xie F, Pu LQ, Magee WP 3rd, Li QF. Autologous Stem Cell Transplantation Promotes Mechanical Stretch Induced Skin Regeneration: A Randomized Phase I/II Clinical Trial. EBioMedicine. 2016 Nov;13:356-364. doi: 10.1016/j.ebiom.2016.09.031. Epub 2016 Oct 1. PMID 27876353